CLINICAL TRIAL: NCT06075186
Title: Assessing Anesthesiologists' Secondary Victim Experience and Quality of Support Resources.
Brief Title: Secondary Victim Awareness of Anesthesiologists
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Faruk Cicekci, principal investigator, Selcuk University
Other Study IDs: farukcicekci7
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Questionnaire
Keywords: Secondary Victim; SVEST scale; Anesthesiologist

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: A survey to assess anesthesiologists' secondary victim experience and quality of support resources. — cross-sectional descriptive questionnaire

SUMMARY:
Every professional working in the medical field may encounter medical errors and patient safety issues during their careers. Wu, et al. He coined the term 'second victim', which was used for the first time in 2000. In a patient safety incident, the patient is the first to be affected, while the second to be affected are the healthcare professionals (physicians, assistants, nurses, and medical staff) who are the potential causes of the incident and who are adversely affected by the consequences of this incident. That is, secondary victims are characterized as healthcare professionals who are involved in unexpected adverse patient events and experience occupational or psychological difficulties. Almost half of healthcare professionals have been reported to experience the second victim phenomenon during their professional careers. Medical errors or adverse events can deeply affect healthcare professionals and have long-term effects, leading to permanent consequences. In the medical field, identifying the origins of errors plays a vital role in preventing future errors. Second victims can encourage constructive change by not only criticizing the healthcare system but also contributing to the improvement of healthcare institutions. Burlison and his team developed and validated a tool they called the "Second Victim Experience and Support Tool" (SVEST) to understand the coping process of second victims and identify necessary support resources. Koca and colleagues conducted a validation study of the translation and psychometric evaluation of the SVEST (T-SVEST) in Turkey. Our study aims to evaluate the secondary victim experience of anesthesiologists and the quality of support resources.

DETAILED DESCRIPTION:
This study will be planned between April 2023 and December 2023 at Selçuk University, Department of Anesthesiology and Reanimation. Physicians who are volunteers and actively working as Anesthesiology and Reanimation Physicians will be included in the study. The study will be conducted as an online survey using demographic data and the T-SVEST scale. Questionnaire; These consist of 3 parts; demographic survey (7 items). Secondary Victim Experience Awareness Survey (29 items) and Secondary Victim Support Option Desirability (7 items). Secondary Victim Experience Awareness Survey and 5-point Likert Scale for Secondary Victim Support Option Desirability were used. The study population consists of 200 Anesthesiology and Reanimation physicians. Svest scale; psychological distress (4 items), physical distress (4 items), colleague support (4 items), supervisor support (4 items), organizational support (3 items), non-work support (2 items), and personal self-efficacy (4 items). It takes into account 7 dimensions: The instrument also assesses 2 outcome variables, intention to change jobs (2 items) and absenteeism (2 items). Moreover; The latter provides a seven-item section as response options for victims to report the forms of support they would like from their organizations. After the survey was presented to the volunteers and the desired sample level was reached, it was planned to use IBM SPSS Statistics Version 27.0.1.0 program to complete the study statistics. Secondary victim experiences and quality of support resources will be compared based on demographic data. All items in the demographic data will be compared for psychological distress, physical distress, peer support, supervisor support, organizational support, non-work support, personal self-efficacy, intention to change jobs, and absenteeism.

ELIGIBILITY:
Inclusion Criteria:

* To be actively working as an Anesthesiology and Reanimation Physician
* Volunteering to participate in the study

Exclusion Criteria:

* Not actively working as an Anesthesiology and Reanimation Physician
* Not volunteering to participate in the study

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be conducted by collecting multicenter data from actively working anesthesiologists.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Secondary victim experience in anesthesiologists | 9 month
  SVEST scale; psychological distress (4 items), physical distress (4 items), colleague support (4 items), supervisor support (4 items), organizational support (3 items), non-work support (2 items), and personal self-efficacy (4 items). It takes into account 7 dimensions: The instrument also assesses 2 outcome variables, intention to change jobs (2 items) and absenteeism (2 items).

SECONDARY OUTCOMES:
Assessing the quality of support resources | 9 month
  The latter provides a seven-item section for victims to report the forms of support they would like from the institutions in which they work.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No